CLINICAL TRIAL: NCT05075109
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Upper Limb Spasticity, Strength and Functional Status in Stroke Patients
Brief Title: TENS and Spasticity in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01037 Komal Mazhar
Record Dates: First submitted 2021-09-17; First posted 2021-10-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Spasticity; Upper limb; TENS
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Frequency TENS (Experimental): high frequency TENS (100 Hz, 200 us) over the muscle belly of triceps and wrist extensors, for 5 days per week over 8 weeks combined with task related training.
  Interventions: Device: High Frequency TENS
- Low Frequency TENS (Experimental): low frequency TENS (20 Hz, 0.2 us) over the muscle belly of triceps and wrist extensors, for 5 days per week over 8 weeks with task related training.
  Interventions: Device: Low Frequency TENS
- Task Related Training (Active Comparator): postural control, shoulder mobilization, weight bearing exercises, functional activities that will comprise of simple tasks to more advanced movement patterns
  Interventions: Other: Task Related Training

INTERVENTIONS:
Device: High Frequency TENS — 30 minutes of high frequency TENS (100 Hz, 200 us) over the muscle belly of triceps and wrist extensors, for 5 days per week over 8 weeks combined with task related training.
  Arms: High Frequency TENS
Device: Low Frequency TENS — 30 minutes of low frequency TENS (20 Hz, 0.2 us) over the muscle belly of triceps and wrist extensors, for 5 days per week over 8 weeks. And combined with 30 minutes of TRT.
  Arms: Low Frequency TENS
Other: Task Related Training — Each session of TRT would include:
  1. postural control, 2. shoulder mobilization, 3. weight bearing exercises 4. Functional activities that will comprise of simple tasks to more advanced movement patterns as follows:
  * Reaching activities
    1. Forward supported reach with cane on tabletop
    2. Reaching against gravity
    3. Reaching overhead with active wrist/hand movements
    4. Dynamic reaching to target e.g. catch a ball
  * Grasping, holding and release
    1. Grasp, hold and release objects with gravity minimized
    2. Pick up and move/release small objects on table
    3. Pick up and move/release large objects without proximal support
    4. Incorporate pinch grips in hold and release including stacking, lifting and overhead activity
  * Upper limb ADL
    1. Brushing hair, putting on scarf
    2. Opening bottles, turning off water tap
    3. Writing, drawing
    4. Folding of towels, hanging towels and setting table
    5. Self-feeding
  Arms: Task Related Training

SUMMARY:
study aims to evaluate the efficacy of high and low frequency TENS on spasticity, strength and functional status in stroke patients. It may provide further knowledge concerning the use of TENS for motor impairments in stroke patients and may clarify ambiguities to some extent.

DETAILED DESCRIPTION:
Despite the positive effects of electrical stimulation proved on motor impairments of affected limb, the evidence is still not conclusive. There still remains a question mark regarding the effectiveness and optimal stimulation parameters of TENS. there has been conflict regarding the TENS parameters (frequency, duration, intensity) among different studies. To date TENS parameters used in different studies to reduce spasticity range from frequency of 1.7-100 Hz, duration from 15-60 minutes and sessions from 1-30. The use of different parameters may account for the contradictory results related to effectiveness of TENS.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female aged 40-70 years
* Middle cerebral artery (MCA) stroke
* 6 months after stroke
* Mini-mental state examination (MMSE)more than 24
* Modified Ashworth scale score between1 and 2

Exclusion Criteria:

* Patients with multiple sclerosis, spinal cord injury or with other pre-existing neurological disorders.
* Patients with orthopedic condition affecting upper extremity
* Patients with contraindication to TENS, like skin damaged etc.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 8 weeks
  Modified Ashworth Scale (MAS) is a subjective method used clinically to measure spasticity. It has verified validity to test spasticity. MAS is six point scale (0,1,2,3,4,5) with a 0 indicating no resistance and 5 indicating rigidity. It has good intra and inter-rater reliability with inter-rater reliability of r= 0.92 and intra-rater reliability at r=0.86.

SECONDARY OUTCOMES:
Manual Muscle Testing (MMT) | 8 weeks
  MMT is used as a clinical procedure to test the strength of muscle. During procedure the therapist observe the muscle's ability to produce movement and respond to manual resistance to assign ordinal scores. 6 point scale is used to grade the muscle strength, (0,1,2,3,4,5) where 0 indicates no perceptible muscle contraction while 5 indicates maximum force generation by muscle against maximum resistance. The MMT has well established validity relative to other measures of muscle strength.
Action Research Arm Test (ARAT) | 8 weeks
  The action research arm test has been used to assess the ability of affected limb to perform activities. It consists of 19 items in which subject is asked to grasp, move and release objects of different shape and size. They are also asked to perform gross movements. Each item is scored on 4 point scale with 0 indicating no action can be performed and 3 indicating that action has been performed successfully within time. validity and reliability of ARA has been confirmed with intra-rater reliability ranging from 0.71-0.99.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Chandka Medical College Hospital, Larkana, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No